CLINICAL TRIAL: NCT04013477
Title: A Single-blinded, Placebo- and Active-controlled, Parallel, Single-ascending Dose Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetics of DA-5207 Transdermal Delivery System in Healthy Adults
Brief Title: Single-ascending Dose Phase 1 Clinical Trial to Evaluate the Safety and PK of DA-5207 TDS in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA5207_ADK_Ia
Record Dates: First submitted 2019-06-26; First posted 2019-07-09 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Healthy
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort1 (Experimental): drug : DA-5207 80mg/40cm²
  placebo : 40cm²
  Interventions: Drug: DA-5207
- Cohort2 (Experimental): drug : DA-5207 120mg/60cm²
  placebo : 60cm²
  Interventions: Drug: DA-5207
- Cohort3 (Experimental): drug : DA-5207 160mg/80cm²
  placebo : 80cm²
  Interventions: Drug: DA-5207
- Cohort4 (Active Comparator): drug : Aricept
  Interventions: Drug: Donepezil Hydrochloride

INTERVENTIONS:
Drug: DA-5207 — DA-5207 Transdermal Delivery System
  Arms: Cohort1; Cohort2; Cohort3
Drug: Donepezil Hydrochloride — donepezil HCl 10mg QD
  Other Names: Aricept
  Arms: Cohort4

SUMMARY:
A single-blinded, placebo- and active-controlled, parallel, single-ascending dose phase 1 clinical trial to evaluate the safety and pharmacokinetics of DA-5207 transdermal delivery system in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Health Male Volunteers (Age : 19~55 years)
* Body Weight : Male≥55kg, Female≥50kg
* 18.5≤BMI<25.0

Exclusion Criteria:

* Galactose intolerance, Lapp lactase deficiency, Glucose-galactose malabsorption
* Allergy or Drug hypersensitivity
* Clinically significant Medical History
* AST, ALT > Upper Normal Range*1.25, eGFR<60mL/min/1.73m²
* Heavy alcohol intake (more than 210g/week)
* Heavy smoker (more than 10 cigarettes/day)
* Heavy caffeine intake

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
AUC | patch : 21days, oral : 11days
  area under the concentration-time curve
Cmax | patch : 21days, oral : 11days
  maximum serum concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Center, Severance Hospital, Seoul, South Korea